CLINICAL TRIAL: NCT07323654
Title: A Phase 2b, Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter, Dose-ranging Study Investigating the Efficacy and Safety Profile of KT-621 Administered Orally to Adult Participants With Uncontrolled Moderate to Severe Eosinophilic Asthma
Brief Title: A Study of KT-621 Administered Orally to Adult Participants With Moderate to Severe Eosinophilic Asthma
Acronym: BREADTH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kymera Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KT621-AS-202
Record Dates: First submitted 2026-01-06; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Eosinophilic Asthma
Keywords: kt-621; stat6 degrader; stat6; targeted protein degrader; Phase 2; phase 2b
MeSH Terms: conditions — Pulmonary Eosinophilia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: KT-621 Dose 1 (Experimental)
  Interventions: Drug: KT-621
- Group 2: KT-621 Dose 2 (Experimental)
  Interventions: Drug: KT-621
- Group 3: KT-621 Dose 3 (Experimental)
  Interventions: Drug: KT-621
- Group 4: Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: KT-621 — Oral drug
  Arms: Group 1: KT-621 Dose 1; Group 2: KT-621 Dose 2; Group 3: KT-621 Dose 3
Other: Placebo — Oral placebo matched to KT-621
  Arms: Group 4: Placebo

SUMMARY:
This Phase 2b study is designed to evaluate the safety and efficacy of KT-621 in participants with uncontrolled moderate to severe eosinophilic asthma.

The main goals of this study are to investigate how effective KT-621 is at treating uncontrolled moderate to severe eosinophilic asthma, the safety and tolerability of KT-621, and how KT-621 behaves in the body.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years old (or the legal age of consent in the jurisdiction in which the study is taking place) to 75 years of age, inclusive, at the time of signing the ICF.
* Must have a physician diagnosis of asthma for at least 1 year prior to the Screening visit.
* Must be on a stable regimen of medium- to high- dose inhaled corticosteroid (ICS), in combination with a long-acting β2-agonist (LABA). The regimen may include additional controller medications used for at least 12 weeks, at a stable dose and regimen, with no change in the dose or frequency of administration for at least 4 weeks prior to the Screening visit and between the Screening and Baseline visits.
* Must have a pre-bronchodilator FEV1 40 to 80% of predicted normal at the Screening and Baseline visits, prior to randomization.
* Must have an ACQ-5 score ≥ 1.5 at the Screening and Baseline visits, prior to randomization.
* Must have a FeNO level of ≥ 25 ppb at the Screening and Baseline visits.
* Must have a demonstrated evidence of reversible airway obstruction by post-bronchodilator (albuterol/salbutamol) reversibility of FEV1 ≥12% and ≥200 mL at Screening.
* Must have an absolute blood eosinophil count must be ≥ 0.30 × 10^9/L at Screening.
* Must have a documented history of at least 1 asthma exacerbation requiring either treatment with systemic corticosteroids (intramuscular, intravenous, or oral) and/or hospitalization or an emergency/urgent medical care visit for acute asthma worsening within the past 52 weeks prior to Screening.
* Must agree to contraceptive requirements in compliance with the clinical study and local requirements.
* Must be willing and able to comply with scheduled visits, treatment plan, laboratory tests, other study-related procedures, and questionnaires, including completing the electronic diary (e-diary), for the duration of the study as required by the study protocol.

Exclusion Criteria:

* Must not have any clinically significant pulmonary disease other than asthma.
* Must not have had an asthma exacerbation, requiring either treatment with systemic corticosteroids (intramuscular, intravenous, or oral) and/or hospitalization or an emergency/urgent medical care visit for acute asthma worsening, at any time from 4 weeks prior to the Screening visit up to and including the Baseline visit.
* Must not have any other clinically significant disease, condition, or medical history that, in the opinion of the Investigator, would interfere with participant safety, study evaluations, and/or study procedures.
* Must not be pregnant or breastfeeding; must not be a woman planning to become pregnant or breastfeed during the study.
* Must not have results from clinical laboratory safety tests that are outside the local reference range at Screening.
* Must not have been dosed with any investigational drug or device in a clinical study within 8 weeks or 5 half-lives (whichever is longer) of KT-621 administration.
* Must not have any known factor, condition, or disease that might interfere with treatment compliance, study conduct or interpretation of the results.
* Must not be a current smoker of nicotine/tobacco as well as non-nicotine products, have a smoking history of ≥ 10 pack years, or use vaping products, including electronic cigarettes. Former smokers with a smoking history of < 10 pack years and users of vaping or e-cigarette products must have stopped for at least 26 weeks prior to the Screening visit.
* Must not have a known sensitivity to any of the components of KT-621.
* Must not be a member of the investigational team or his/her immediate family.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in pre-bronchodilator FEV1 | From baseline to Week 12

SECONDARY OUTCOMES:
Change from baseline in post-bronchodilator FEV1 | From baseline to Week 12
Change from baseline in Asthma Control Questionnaire 5-question version (ACQ-5) score | From baseline to Week 12
Change from baseline in Standardized Asthma Quality of Life Questionnaire [AQLQ(S)] Global Score | From baseline to Week 12
Incidence of treatment-emergent adverse events (TEAEs) | From baseline through Week 16
Incidence of treatment-emergent serious adverse events (SAEs) | From baseline through Week 16
Plasma concentration of KT-621 derived from plasma concentration time data | From baseline to Week 16

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Kymera Investigative Site, Tampa, Florida
  - Kymera Investigative Site, Edmond, Oklahoma

IPD SHARING:
Plan to Share IPD: No